CLINICAL TRIAL: NCT04067765
Title: Using Neuroeconomics to Characterize State-Based Increases and Decreases in Alcohol Value
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: R01AA027255-01A1 (NIH)
Record Dates: First submitted 2019-08-16; First posted 2019-08-26 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder; Alcohol Drinking
Keywords: Alcohol; Neuroeconomics; Demand; Cues
MeSH Terms: conditions — Alcoholism; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Participants will undergo a validated cue exposure protocol involving exposure to neutral beverage cues followed by exposure to alcohol beverage cues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neutral Cue, then Alcohol Cue (Experimental): Participants first completed an in-scanner neutral cue exposure prior to the first two in-scanner alcohol purchase tasks runs. Participants then received an in-scanner alcohol cue exposure prior to the final two in-scanner alcohol purchase task runs. Cue exposures consisted of images of neutral (water) or alcohol (beer, wine, liquor) beverages and an imaginal script describing a drinking scenario.
  Interventions: Behavioral: Cue Exposure

INTERVENTIONS:
Behavioral: Cue Exposure — Participants will undergo a validated in-scanner alcohol cue and neutral cue exposure protocol involving passive viewing of images of alcohol beverages (beer, wine, or liquor) and neutral beverages (water).

SUMMARY:
This study uses techniques from an area of research known as neuroeconomics, which integrates concepts and methods from psychology, neuroscience, and economics to better understand how people make decisions and how these decisions are supported by the brain. One neuroeconomic concept that is especially relevant in the area of addictions is substance demand, or how consumption of a commodity (e.g., alcohol, tobacco, or drugs) is influenced by price and other factors. Previous studies have shown that alcohol demand is related to severity of alcohol misuse, drinking quantity/frequency, and treatment outcomes. In addition, we know that alcohol demand can also fluctuate in response to environmental cues such as alcohol-related stimuli or external contingencies such as important responsibilities the following day. These increase and decreases in consumption and value are clinically significant because they help us understand how people with alcohol use disorders are able to successfully or unsuccessfully modulate their drinking behaviors. This study is examining how the brain responds in these situations and whether these responses differ as a function of severity of alcohol misuse. This study will use functional magnetic resonance imaging (fMRI) to understand brain activity patterns associated with changes in the value of alcohol in the presence of alcohol-related beverage cues relative to neutral-related beverage cue. Participants will be non-treatment-seeking adult heavy drinkers who are recruited from the community to participate in an fMRI scan. During the scan, participants will make decisions about how many alcohol beverages they would consume (hypothetically) at various prices while their brain activity during those decisions is measured. The experimental manipulation involves an in-scanner alcohol cue exposure task in which the drinking decisions will be made after viewing high-quality images of alcoholic (beer/wine/liquor) beverages or neutral (water/juice/soft drinks) beverages.

DETAILED DESCRIPTION:
Neuroeconomics integrates concepts and methods from psychology, economics, and cognitive neuroscience to understand the neurobiological foundations of decision making, and has been increasingly applied to understanding alcohol use disorder (AUD). A novel application of neuroeconomics is the study of alcohol demand, or the value of alcohol as measured by cost-benefit preferences. Alcohol demand paradigms have considerable ecological validity by measuring the impact of internal and external influences on alcohol decision-making, such as price, environmental cues, affective states, or external contingencies. Behaviorally, alcohol demand is elevated among individuals with higher levels of alcohol misuse and predicts treatment response. Alcohol demand also exhibits state-like properties, including increases following exposure to alcohol-related cues. The overall goal of the proposed studies is to characterize the neural activity that subserves these established behavioral findings using a novel functional MRI paradigm.

The primary aim is to examine the patterns of neural activation underlying increases in the value of alcohol in response to alcohol cues. The study will use a within-subjects design to identify differences in neural activity associated with demand decisions following a validated in-scanner cue exposure protocol consisting of exposure to neutral beverage cues and exposure to alcohol beverage cues in a sample of adult heavy drinkers.

Using a novel neuroeconomics approach, this study combines a highly ecologically-valid alcohol demand paradigm with an experimental manipulation that models clinically-relevant influences on drinking decisions. Studying these contextual influences may help clarify the neural signatures that underlie drinking moderation vs. unconstrained drinking, and how these processes are impacted by AUD. If successful, this study will provide a foundation for examining neural predictors of successful recovery or response to treatment vs. relapse. More broadly, findings from this study have high potential to significantly enhance the clinical relevance of alcohol neuroscience.

ELIGIBILITY:
Inclusion Criteria:

* 21-55 years old;
* Right-handed;
* Fluent English speaker;
* Heavy drinker (i.e., on average > 14/7 drinks per week for males/females in past three months;
* Average of 1 heavy drinking episode weekly (heavy drinking episode = 5+/4+ for males/females) over past three months

Exclusion Criteria:

* Currently receiving treatment, or seeking treatment, for alcohol related problems;
* Current Diagnostic and Statistical Manual (DSM-5) substance use disorder other than alcohol or tobacco;
* Weekly or more frequent use of recreational drugs;
* History of schizophrenia-spectrum disorders, psychotic disorders, bipolar disorder, or PTSD;
* History of neurocognitive disorder or impairment;
* MRI contraindications (e.g., metal in body, history of seizure, etc.);
* History of serious brain injury;
* Currently taking psychotropic medications or medications that could affect cerebral blood flow;
* Pregnancy (females);
* Attending any study session with a positive breath alcohol concentration (BrAC > 0.00g%)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Amlung, PhD, Principal Investigator — University of Kansas
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cue Exposure: Within subjects assignment to receive complete both an alcohol cue exposure and neutral cue exposure in a sequential order (neutral followed by alcohol cues. Each run was preceded by a slideshow of pictures of neutral or alcohol beverages. Following standard practice in laboratory cue exposure paradigms, the neutral cues were presented first (prior to runs 1-2) followed by the alcohol cues (prior to runs 3-4) to minimize potential of carryover effects. Neutral cues depicted various water beverages and alcohol cues depicted the participant's preferred alcohol type (beer, wine, or liquor). Each exposure included 30 cues presented for 3s each. Prior to the first neutral and alcohol cue run, an imaginal cue script was read aloud to the participant.
Period: Neutral Cue Exposure (5 Minutes Total)
Arm/Group | Cue Exposure
Started | 72
Completed | 72
Not Completed | 0
Period: Alcohol Cue Exposure (5 Minutes Total)
Arm/Group | Cue Exposure
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Alcohol Cue Exposure: Within subjects assignment to receive complete both an alcohol cue exposure and neutral cue exposure in a sequential order.
Arm/Group | Alcohol Cue Exposure
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants] — Diagnostic Assessment Research Tool (DART) DSM-5 Alcohol Use Disorder
  Participants
    <=18 years | 0
    Between 18 and 65 years | 72
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 67
  More than one race | 5
  Unknown or Not Reported | 0
Alcohol Use Disorders Identification Test (AUDIT) [Mean (Standard Deviation); unit: units on a scale] — The Alcohol Use Disorders Identification Test is a 10-item screening questionnaire assessing quantity/frequency of alcohol consumption and alcohol-related problems experienced over the last 12 months. All items are summed to generate a total AUDIT score, with scores ranging from 0-40. Higher scores representing greater alcohol use disorder severity.
  units on a scale | 12.0 (5.4)
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 0
Education [Mean (Standard Deviation); unit: Years] — Years of Education
  Years | 16.3 (2.0)
Daily Drinking Questionnaire (DDQ) [Mean (Standard Deviation); unit: Drinks/week] — Drinks per week calculated from Daily Drinking Questionnaire
  Drinks/week | 22.3 (13.1)
Diagnostic Assessment Research Tool (DART) for DSM-5 Alcohol Use Disorder [Count of Participants; unit: Participants] — Semi-structured clinical interview assessing DSM-5 alcohol use disorder diagnoses. Participants received a diagnosis of alcohol use disorder if they endorsed 2 or more criteria on the DART interview. Variable reflects the count of participants meeting DSM-5 criteria for alcohol use disorder.
  Participants | 49
30 Day Timeline Follow-Back Interview [Mean (Standard Deviation); unit: Drinks/week] — Drinks per week calculated from 30-day alcohol timeline follow-back interview
  Drinks/week | 20.3 (12.9)

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Demand Intensity
Description: Intensity is defined as the self-consumption in standard drinks at free price. Participants could select between 0-10 standard sized alcohol drinks on the in-scanner alcohol purchase task paradigm. The mean intensity was calculated separately for the two neutral cue runs and the two alcohol cue runs.
Time Frame: Collected during each of 4 runs of the FMRI Alcohol Purchase Task. Duration of each run was approximately 6 minutes and included 26 trials.
Measure: Mean (Standard Error); unit: Drinks
Arm/Group | Alcohol Cue Exposure
Number analyzed (Participants) | 72
Drinks
  Neutral Cue Exposure | 7.42 (0.30)
  Alcohol Cue Exposure | 7.85 (0.27)

2. Primary Outcome: Alcohol Demand Breakpoint
Description: Breakpoint is defined as the first price on the alcohol purchase task that suppressed consumption to zero drinks. The mean breakpoint was calculated separately for the two neutral cue runs and the two alcohol cue runs.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Dollars
Arm/Group | Alcohol Cue Exposure
Number analyzed (Participants) | 68
Dollars
  Neutral Cue Exposure | 28.77 (1.67)
  Alcohol Cue Exposure | 32.48 (1.45)

3. Primary Outcome: Alcohol Demand Omax
Description: Omax is defined as the maximum total expenditure on alcohol for the in-scanner alcohol purchase task. The mean Omax was calculated separately for the two neutral cue runs and the two alcohol cue runs.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Dollars
Arm/Group | Alcohol Cue Exposure
Number analyzed (Participants) | 72
Dollars
  Neutral Cue Exposure | 49.54 (6.32)
  Alcohol Cue Exposure | 60.63 (8.39)

4. Primary Outcome: Alcohol Demand Elasticity
Description: Elasticity is defined as the change in consumption (in drinks) as a function of increases in price per drink (in dollars). This index was modeled using an exponentiated demand curve model as reported in [Koffarnus, M. N., Franck, C. T., Stein, J. S., & Bickel, W. K. (2015). A modified exponential behavioral economic demand model to better describe consumption data. Experimental and clinical psychopharmacology, 23(6), 504-512. https://doi.org/10.1037/pha0000045]. This nonlinear model generates a best fitting value for an alpha parameter, reflecting the rate of change in elasticity over increasing price. Higher alpha values reflect greater elasticity (greater sensitivity in consumption with increases in price). There is no theoretical range as this is a free parameter in the model. Mean alpha values were calculated separately for the two neutral cue runs and the two alcohol cue runs.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: drinks consumed/price (dollars)
Arm/Group | Alcohol Cue Exposure
Number analyzed (Participants) | 72
drinks consumed/price (dollars)
  Neutral Cue Exposure | 0.006 (0.001)
  Alcohol Cue Exposure | 0.003 (0.001)

5. Secondary Outcome: Alcohol Craving
Description: Subjective alcohol craving was assessed using three 100-point scales, including how much they want alcohol, crave alcohol, and their urge for alcohol. A score of 0 indicates the lowest level of craving; a score of 100 indicates the highest amount of craving. The three items were averaged into a composite craving score.
Time Frame: Collected immediately after the first neutral cue exposure and immediately after the first alcohol cue exposure.
Measure: Mean (Standard Error); unit: Points
Arm/Group | Alcohol Cue Exposure
Number analyzed (Participants) | 72
Points
  neutral cue exposure | 19.72 (2.49)
  alcohol cue exposure | 27.99 (2.84)

ADVERSE EVENTS:
Time Frame: Baseline visit to MRI scan visit. Median time frame = 23 days (minimum time frame 2 days; maximum time frame 88 days)
Description: Standard definition of adverse event and serious adverse event were used.
Groups:
- Neutral Cue Exposure: Neutral cue exposure during fMRI scan
- Alcohol Cue Exposure: Alcohol cue exposure during fMRI scan
Arm/Group | Neutral Cue Exposure | Alcohol Cue Exposure
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 0/72 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT04067765/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT04067765/SAP_001.pdf
  • Informed Consent Form (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT04067765/ICF_002.pdf